CLINICAL TRIAL: NCT05096637
Title: PreventiPlaque - Digital Secondary Prevention in Cardiovascular Disease to Improve Therapy Adherence
Brief Title: Digital Secondary Prevention in Cardiovascular Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Julia Lortz, PD Dr. med., University Hospital, Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20-9157-BO
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Atherosclerotic Plaque
MeSH Terms: conditions — Plaque, Atherosclerotic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Patients receive the best medical care according to current guideline recommendations without access to the app
- intervention group (Experimental): Patients receive the best medical care according to current guideline recommendations with full access to the app. This includes access to relevant findings including ultrasound images of the carotid artery, lipid profile, blood pressure values, and weight.
  Interventions: Other: PreventiPlaque App

INTERVENTIONS:
Other: PreventiPlaque App — PreventiPlaque is an app that supports patients with atherosclerotic plaque by strengthening their adherence.
  Arms: intervention group

SUMMARY:
Although advances in knowledge of the prevention, diagnosis and treatment of atherothrombosis are encouraging, cardiovascular diseases (CVD), with acute and chronic ischemic heart disease in particular, remain a major cause of disability and premature death throughout the world.

Cardiac rehabilitation (CR) and secondary prevention are coordinated multidimensional evidence-based strategies that aim to assist patients with acute and chronic ischemic heart disease return to an active and satisfying life and to prevent the recurrence of further cardiac events. Since CR is time limited after an acute event, secondary prevention proposes a continuum where care is provided for the rest of a person's life according to the existence of cardiovascular risk factors. Secondary prophylaxis is fundamental for the recovery of the patient, but in most cases, it is only insufficiently implemented.

To ensure adequate resources for the delivery of health care and to further improve the level of care, care-delivery models need to be changed in a way that patients themselves become more involved in their own care. Mobile health (mHealth) is a rapidly growing health delivery methodology with the potential to impact on health care research, health care delivery and health outcomes.

Therefore, the aim of the study is to determine the impact of plaque visualization using a digital intervention on treatment adherence to improve the cardiovascular risk profile. Participants will be randomized into two groups: intervention group and control group. Participants of the control group receive the best medical care according to current guideline recommendations without access to the app. Participants of the intervention group receive the best medical care according to current guideline recommendations with full access to the Smartphone application at time of study begin until the completion of the follow-up period of 12 months. The access to the app includes access to relevant findings including ultrasound images of the carotid artery, lipid profile, blood pressure values, and weight.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound evidence of atherosclerotic plaque in one or both carotid arteries
* Own a smartphone and know how to use apps
* presumed life expectancy of more than one year
* willing to comply with the protocol and provide written informed consent

Exclusion Criteria:

* congestive heart failure with NYHA (New York Heart Association classification) III-IV symptoms
* severe valve disease
* no german knowledge
* unwillingness to user the app and/or undergo diagnostic procedures

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Change in cardiovascular risk profile | baseline, 3 months follow-up, 6 months follow-up, 9 month follow-up, end of study after 12 months
  Measured via SCORE2 (Systematic Coronary Risk Evaluation) risk calculator

SECONDARY OUTCOMES:
Change in LifeSimple7-Score | baseline, 3 months follow-up, 6 months follow-up, 9 month follow-up, end of study after 12 months
  Measured by Score released by the American Heart Association (AHA)
Change in LDL-cholesterol | baseline, 3 months follow-up, 6 months follow-up, 9 month follow-up, end of study after 12 months
  measured in mg/dl
Change in body weight | baseline, 3 months follow-up, 6 months follow-up, 9 month follow-up, end of study after 12 months
  measured in kg
Change in blood pressure | baseline, 3 months follow-up, 6 months follow-up, 9 month follow-up, end of study after 12 months
  measured in mmHg
Reported physical activity | baseline, 3 months follow-up, 6 months follow-up, 9 month follow-up, end of study after 12 months
  measured via self-report question
Change in cigarette dependency | baseline, 3 months follow-up, 6 months follow-up, 9 month follow-up, end of study after 12 months
  asses via Fagerstrom Test for Cigarette Dependence
Change in reported medication adherence | baseline, 3 months follow-up, 6 months follow-up, 9 month follow-up, end of study after 12 months
  assessed via self-report question
Satisfaction with outpatient care | baseline, 3 months follow-up, 6 months follow-up, 9 month follow-up, end of study after 12 months
  assessed via questionnaire "Satisfaction in outpatient care)

OTHER OUTCOMES:
Patient-centered evaluation of the intervention-app | end of study after 12 months
  assessed via Mobile Application Rating Scale: user version (uMARS)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ullrich G, Bauerle A, Jahre LM, Paldan K, Rosemeyer J, Kalaitzidis C, Rammos C, Teufel M, Rassaf T, Lortz J. Impact of visual presentation of atherosclerotic carotid plaque on cardiovascular risk profile using mHealth technologies. NPJ Digit Med. 2025 Jan 22;8(1):47. doi: 10.1038/s41746-024-01423-y. PMID 39843925